CLINICAL TRIAL: NCT01194154
Title: A Randomized Controlled, Single-blind, Proof-of-concept-study to Investigate the Protective Effects of Early Treatment With C.E.R.A. in Patients With Chronic Kidney Disease on Renal Disease Progression (PRIMAVERA-Study)
Brief Title: A Study of Methoxy Polyethylene Glycol-epoetin Beta (Mircera) in Participants With Chronic Kidney Disease (PRIMAVERA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ML22916; 2009-015114-22
Record Dates: First submitted 2010-08-25; First posted 2010-09-02 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Mircera (Experimental)
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta — Methoxy polyethylene glycol-epoetin beta 30 microgram (mcg) subcutaneous injection once monthly up to 24 months with sequential dose adjustments to 50 mcg or 75 mcg depending on change of hemoglobin values of more than 1.0 gram (g)/ deciliter (dL).
  Other Names: Mircera, C.E.R.A.
  Arms: Mircera
Drug: Placebo — Placebo matching to Methoxy polyethylene glycol-epoetin beta subcutaneous injection once monthly up to 24 months.
  Arms: Placebo

SUMMARY:
This randomized, single-blind, proof-of-concept study will investigate the protective effects of early treatment with Mircera in participants with chronic kidney disease on renal disease progression. Participants will be randomly assigned to receive 30 microgram (mcg) Mircera as subcutaneous injection once monthly or matching placebo. Depending on change of hemoglobin values, the dose of Mircera can be adjusted to 50 mcg or 75 mcg once monthly. The anticipated time on study treatment is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* For diabetic participants: Type 2 diabetes mellitus with glycated hemoglobin (HbA1c) greater than (>) 7% or anti-diabetic treatment
* For renal allograft recipients: Status at least 6 months post transplantation
* Chronic kidney disease stage III
* Urinary albumin-to-creatinine ratio less than (<) 3000 milligram (mg)/gram (g) or total protein <3000 mg/ 24 hour urine sample where applicable

Exclusion Criteria:

* Hemoglobin-level < 11 or > 14 g/deciliter (dL)
* Average systolic blood pressure (SBP) > 140 millimeter of mercury (mm Hg) or average diastolic blood pressure (DBP) > 90 mm Hg
* Initiation of angiotensin converting enzyme inhibitor, angiotensin 2 receptor blocker or aliskiren treatment less than 3 months before enrolment
* Present and known iron deficiency
* HbA1c >9%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- Germany (33):
  - Uniklinik RWTH Aachen; Med. Klinik II; Klinik für Nephrologie und klinische Immunologie, Aachen
  - Dialysepraxis Dr. Stallforth, Dr. Kirschner, Dr. Al-Sarraf und Dr. Pawlik, Augsburg
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V. im Kurhaus, Bad König
  - Charité - Klinikum Mitte; Medizinische Klinik Für Nephrologie, Berlin
  - Charité - Campus Benjamin Franklin; Zentrum fuer Innere Medizin, Med. Klinik I, Berlin
  - Gemeinschaftspraxis Dres. Erika Eger, Frank Seibt, Oliver Eike u.w. - Dialysezentrum Treptower Park, Berlin
  - Dialyse-Institut Bovenden, Bovenden
  - Kliniken der Stadt Köln gGmbH Krankenhaus Merheim, Cologne
  - Universitätsklinikum "Carl Gustav Carus"; Medizinische Klinik III, Dresden
  - DaVita Clinical Research Deutschland GmbH, Düsseldorf
  - Universitätsklinikum Essen Zentrum f.Innere Medizin Abt.Nephrologie, Essen
  - Klinik Johann Wolfgang von Goethe Uni; Zentrum der Inneren Medizin; Medizinische Klinik III, Frankfurt
  - Uniklinikum Heidelberg, Heidelberg
  - Dialysepraxis Prof.Dr.med. Michael Rambausek Dres. Stephan Matthias und Gabriele Kunowski - Dialysz., Heilbronn
  - Nephrologisches Zentrum Hilden am St. Josefs-Krankenhaus, Hilden
  - Universitaetsklinikum des Saarlandes; Klinik f. Innere Medizin IV, Homburg/Saar
  - Dres. Jan Nawka und Frank Pistrosch, Hoyerswerda
  - Westpfalz-Klinikum Gmbh; Nephrologie/Transplantationsmedizin, Kaiserslautern
  - PHV Patienten-Heimversorgung Dialyse-Station, Kiel
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck, Med. Klinik I, Transplantationszentrum, Lübeck
  - Gemienschaftspraxis Dres. Leistikow, Rachti & Sandner, Mannheim
  - Dres. Michael Koch Hannelore Klimke Wolfgang Kulas u.w., Mettmann
  - Klinikum Innenstadt Medizinische Klinik; Abt.Endokrinologie und Diabetologie, München
  - Klinikum d.Universität München Campus Großhadern, München
  - Nierenzentrum Bogenhausen/Perlach; Praxis für Nierenheilkunde, München-Bogenhausen
  - Universitätsklinikum Münster Innere Medizin D, Münster
  - Dres. Georg Fuchs und Nexhat Miftari, Neckarsulm
  - Nephrologische Praxis Neunkirchen - Dr.med. Klemens Dorr und Artem Goldmann, Neunkirchen/Saar
  - Dialysezentrum Saarlouis, Saarlouis
  - Gemeinschaftspraxis Rosemarie Krämer und Lars Rothermund, Ulm
  - Nephrologisches Zentrum, Velbert
  - Nephrologisches Zentrum Dialyse-Institut, Villingen-Schwenningen
  - KfH Kuratiorium für Dialyse und Nierentransplantation e.V., Wiesbaden

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 241 participants were enrolled, 2 participants in the Mircera group and 4 participants in the placebo group did not receive medication.
Groups:
- Mircera: Methoxy polyethylene glycol-epoetin beta 30 microgram (mcg) subcutaneous injection once monthly up to 24 months with sequential dose adjustments to 50 mcg or 75 mcg depending on change of hemoglobin values of more than 1.0 gram (g)/ deciliter (dL).
Period: Overall Study
Arm/Group | Mircera | Placebo
Started | 117 | 124
Full Analysis Set | 115 | 120
Safety Analysis Set | 118 (3 participants randomized to placebo but received MIRCERA and included in MIRCERA arm (as treated).) | 117 (3 participants randomized to placebo but received MIRCERA and included in MIRCERA arm (as treated).)
Completed | 68 | 91
Not Completed | 49 | 33
Not completed — Adverse Event | 12 | 7
Not completed — Lost to Follow-up | 2 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Blood pressure increase | 5 | 3
Not completed — Hemoglobin decrease | 0 | 1
Not completed — Hemoglobin increase | 12 | 3
Not completed — Skipping of CERA treatment at two visits | 3 | 0
Not completed — Treatment with prohibited medication | 4 | 5
Not completed — Other | 4 | 0
Not completed — Did not receive study medication | 2 | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomized participants who received at least one dose of the study medication and provided any successive estimated glomerular filtration rate (eGFR) measurement.
Groups:
- Mircera: Methoxy polyethylene glycol-epoetin beta 30 mcg subcutaneous injection once monthly up to 24 months with sequential dose adjustments to 50 mcg or 75 mcg depending on change of hemoglobin values of more than 1.0 g/dL.
- Total: Total of all reporting groups
Arm/Group | Mircera | Placebo | Total
Number analyzed (Participants) | 115 | 120 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.37 (12.26) | 62.97 (14.30) | 63.17 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 71 | 76 | 147

OUTCOME MEASURES:

1. Primary Outcome: Yearly Reduction Rate of Estimated Glomerular Filtration Rate (eGFR) Calculated by Modification of Diet in Renal Disease With 4 Variables (MDRD-4)
Description: The yearly reduction in eGFR was calculated using the MDRD-4 formula. This formula is based on age, sex, and serum creatinine and eGFR values are calculated as follows: GFR in milliliter per minute (mL/min) per 1.73 meter square (m^2) = 175 x Serum Cr^-1.154 x age^-0.203 x 0.742 (if female). The yearly reduction rate (mL/min/1.73m^2 / Year) is defined as -365.25 multiplied by Beta, where Beta is the slope parameter derived for each participants separately by simple linear regression of the change from baseline in participant's eGFR measurements (from Baseline to Visit 24) on the actual day of measurement.
Time Frame: 24 months
Population: FAS included all randomized participants who received at least one dose of the study medication and provided any successive eGFR measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m^2/year
Arm/Group | Mircera | Placebo
Number analyzed (Participants) | 115 | 120
mL/min/1.73m^2/year | 3.04 [1.20 to 4.87] | 0.82 [-0.96 to 2.61]
Statistical Analysis 1: Comparison: Mircera vs Placebo; Test type: Superiority or Other; p = 0.657, Wilcoxon (Mann-Whitney); treatment effect = 2.21, 95% CI 2-sided [-0.35 to 4.78] — An analysis of covariance (ANCOVA) model with adjustment for baseline eGFR was used to obtain an estimate of the treatment difference

2. Secondary Outcome: Yearly Reduction Rate of Estimated Glomerular Filtration Rate (eGFR) Calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
Description: The eGFR value calculated using the CKD-EPI equation. The formula used is based on age, sex, ethnicity, and serum creatinine and eGFR values are calculated as follows: GFR in mL/min per 1.73 m^2 = 141 x min (SerumCr/k; 1)^a x max(SerumCr/k; 1)^(-1.209) x 0.993^age x F x B, where k=0.7 for female (else=0.9); a=-0.329 for female (else=-0.411), F=1.018 for female (else=1), B=1.159 for black (else=1), min/max=minimum/maximum of listed values. The Yearly Reduction Rate (mL/min/1.73m^2 / Year) is defined as -365.25 x Beta, where Beta is the slope parameter derived for each participant separately by simple linear regression of the change from baseline in participant's eGFR measurements (from Baseline to Visit 24) on the actual day of measurement.
Time Frame: 24 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m^2/year
Arm/Group | Mircera | Placebo
Number analyzed (Participants) | 115 | 120
mL/min/1.73m^2/year | 3.02 [1.03 to 5.00] | 0.78 [-1.16 to 2.72]
Statistical Analysis 1: Comparison: Mircera vs Placebo; Test type: Superiority or Other; p = 0.709, Wilcoxon (Mann-Whitney); treatment effect = 2.24, 95% CI 2-sided [-0.54 to 5.01] — ANCOVA model with adjustment for baseline eGFR was used to obtain an estimate of the treatment difference

3. Secondary Outcome: Change From Baseline in Calculated Creatinine Clearance (Cockcroft-Gault Equation) at Month 24
Description: Creatinine clearance was calculated according to the Cockcroft and Gault Formula. It measures rate creatinine (substance formed from metabolism of creatine) is cleared from blood by kidneys. Normal adult creatinine clearance is greater than or equal to (>=) 90 mL/min. Change from baseline=CC at Week X minus CC at baseline where higher scores represented improved renal function.
Time Frame: Baseline, Month 24
Population: FAS included all randomized participants who received at least one dose of the study medication and provided any successive eGFR measurement. Here, n=number of participants evaluable for each category.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Mircera | Placebo
Number analyzed (Participants) | 115 | 120
mL/min
  Baseline (n=115, 120) | 53.18 (15.95) | 52.48 (16.04)
  Change at Month 24 (n=67, 91) | -2.97 (10.52) | -2.08 (9.72)

4. Secondary Outcome: Change From Baseline in Serum Creatinine Concentration at Month 24
Description: Serum creatinine is an indicator of kidney function. Creatinine is a substance formed from the metabolism of creatine, commonly found in blood, urine, and muscle tissue. It is removed from the blood by the kidneys and excreted in urine. Normal adult blood levels of creatinine=45 to 90 micromoles per liter (mcmol/L) for females, 60 to 110 mcmol/L for males, however normal values are age-dependent.
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Mircera | Placebo
Number analyzed (Participants) | 115 | 120
mcmol/L
  Baseline (n=115, 120) | 147.8 (31.71) | 149.3 (35.67)
  Change at Month 24 (n=68, 91) | 7.04 (27.23) | 4.04 (30.99)

5. Secondary Outcome: Change From Baseline in Urinary Albumin Creatinine Ratio (UACR) at Month 24
Description: UACR is defined as the ratio: milligram of albumin per gram of creatinine. The presence of albumin in the urine (macroalbuminuria) is a marker of kidney disease. Albumin and creatinine concentrations were obtained from spot urine samples.
Time Frame: Baseline, Month 24
Population: FAS included all randomized participants who received at least one dose of the study medication and provided any successive eGFR measurement. Number of Participants Analyzed (N) = number of participants evaluable and available with valid data for this outcome measure. Here, n=number of participants evaluable for each category.
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Mircera | Placebo
Number analyzed (Participants) | 110 | 107
mg/g
  Baseline (n=110, 107) | 261.1 (564.0) | 237.3 (699.6)
  Change at Month 24 (n=43, 53) | 173.8 (573.3) | 70.59 (546.8)

6. Secondary Outcome: Change From Baseline in Serum Cystatin C Concentration at Month 24
Description: Cystatin C is a protein which is mainly used as a biomarker of kidney function. If kidney function and GFR decline, the blood levels of cystatin C rise.
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Mircera: Methoxy polyethylene glycol-epoetin beta 30 mcg subcutaneous injection once monthly up to 24 months with sequential dose adjustments to 50 mcg or 75 mcg depending on change of hemoglobin values of more than 1.0 g/ dL.
Arm/Group | Mircera | Placebo
Number analyzed (Participants) | 115 | 120
mg/L
  Baseline (n=115, 120) | 1.79 (0.39) | 1.76 (0.46)
  Change at Month 24 (n=67, 91) | 0.10 (0.29) | 0.02 (0.33)

7. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability or incapacity; and congenital anomaly. Percentage of participants with AEs included participants affected with both SAEs and non-SAEs.
Time Frame: 24 months
Population: The Safety Analysis Set (SAF) included all participants who received at least one dose of study medication. Analysis for SAF was performed according to the study medication actually received (as treated population). Number of participants analyzed=participants evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera | Placebo
Number analyzed (Participants) | 118 | 117
percentage of participants
  SAEs | 35.6 | 41.0
  AEs | 84.7 | 86.3

ADVERSE EVENTS:
Time Frame: 24 months
Description: The Safety Analysis Set (SAF) included all participants who received at least one dose of the study medication. Analysis for SAF was performed according to the study medication actually received ('as treated' population).
Arm/Group | Mircera | Placebo
Serious Adverse Events (participants affected / at risk) | 42/118 | 48/117
Other Adverse Events (participants affected / at risk) | 95/118 | 99/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=118) | Placebo (N=117)
Bronchopneumonia (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 2 | 0
Anal abscess (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 2
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Postrenal failure (Renal and urinary disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Ectropion (Eye disorders) | 1 | 0
Lens dislocation (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Liver disorder (Hepatobiliary disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Tibial torsion (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Aortic anastomosis (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=118) | Placebo (N=117)
Bronchitis (Infections and infestations) | 0 | 9
Influenza (Infections and infestations) | 9 | 9
Nasopharyngitis (Infections and infestations) | 29 | 24
Urinary tract infection (Infections and infestations) | 12 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 8
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 11 | 13
Nausea (Gastrointestinal disorders) | 0 | 8
Oedema peripheral (General disorders) | 11 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 10
Hypertension (Vascular disorders) | 11 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.